CLINICAL TRIAL: NCT00357552
Title: A Pilot Study of Lopinavir/Ritonavir in Participants Experiencing Virologic Relapse on NNRTI-Containing Regimens
Brief Title: Safety and Effectiveness of Lopinavir/Ritonavir in Individuals Who Have Failed Prior HIV Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5230; 1U01AI068636 (NIH)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LPV/r monotherapy (Experimental): Participants will receive lopinavir/ritonavir twice daily for up to 104 weeks. Upon confirmation of virologic failure, emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) once a day will be added to their regimen.
  Interventions: Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir disoproxil fumarate — Once daily
  Other Names: Truvada
Drug: Lopinavir/Ritonavir — Twice daily
  Other Names: Kaletra, Aluvia

SUMMARY:
Most anti-HIV regimens include a non-nucleoside reverse transcriptase inhibitor (NNRTI); however, some individuals fail on these regimens. The purpose of this study is to evaluate the safety and effectiveness of the protease inhibitor (PI) lopinavir/ritonavir (LPV/r) in HIV infected individuals who are failing an anti-HIV regimen that includes an NNRTI.

DETAILED DESCRIPTION:
Standard effective antiretroviral therapy for HIV infected individuals includes three-drug combinations of two nucleoside reverse transcriptase inhibitors (NRTIs) with either a PI or an NNRTI. However, three-drug regimens may not be ideal in resource-limited settings, where viral load and resistance testing may not be readily available. The purpose of this study is to evaluate the safety and efficacy of the PI LPV/r alone in treatment-experienced, PI-naive HIV infected individuals who are experiencing virologic failure on three-drug regimens.

This study will last 104 weeks. All participants will receive LPV/r twice daily for up to 104 weeks. Participants who experience virologic failure will receive emtricitabine/tenofovir disoproxil fumarate once daily in addition to LPV/r twice daily for the remainder of the study.

There will be 16 study visits for participants on LPV/r monotherapy and 12 study visits for participants who have intensified LPV/r with emtricitabine/tenofovir disoproxil fumarate. Blood collection and clinical assessment will occur at all visits; urine collection and resistance testing will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria for Step 1 Participants:

* HIV infected
* Continuous treatment with a three-drug, NNRTI-containing regimen for at least 6 months prior to study entry
* Viral load of 1,000 copies/ml or greater and less or equal to 200,000 copies/ml obtained within 30 days of study entry
* Negative pregnancy test within 48 hours of study entry
* Willing to use acceptable forms of contraception for the duration of the study
* Laboratory values obtained within 30 days of study entry:

  * Hemoglobin greater or equal to 8.0 g/dL
  * Platelet count greater or equal to 50,000/mm3
  * Estimated Creatinine Clearance greater or equal to 60 mL/min x ULN
  * AST (SGOT), ALT (SGPT) and alkaline phosphatase < 3 x ULN
  * Total bilirubin less or equal to 2.5 x ULN
* Ability and willingness of participant or legal guardian/representative to give informed consent

Inclusion Criteria for Step 2 Participants:

* Virologic failure on LPV/r monotherapy defined as viral load of 400 copies/ml or greater after 24 consecutive weeks on LPV/r monotherapy OR virologic failure after initial viral suppression on LPV/r monotherapy
* Estimated creatinine clearance of 60 ml/min or greater
* Negative pregnancy test within 48 hours of entry into Step 2
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria for All Participants:

* Breastfeeding
* Known allergy or sensitivity to study drugs
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with study adherence to study requirements
* History of chronic hepatitis B infection

Exclusion Criteria for Step I Participants:

* Prior use of any protease inhibitor treatment
* Acute therapy for any serious medical condition within 14 days of study entry. For ongoing or chronic therapy, the participant must be on the treatment regimen for at least 14 days, and clinically stable prior to entry. If a potential participant has TB and has received treatment for more than 2 weeks, the TB treatment would have to be modified to include a rifabutin-containing regimen. TB compatible syndromes will also be carefully evaluated prior to entry.

Exclusion Criteria for Step 2 Participants:

- Active opportunistic infection, including tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagalingeswaran Kumarasamy, MBBS, PhD, Study Chair — Y. R. Gaitonde Centre for AIDS Research and Education; John Bartlett, MD, Study Chair — Division of Infectious Diseases, Duke University Medical Center
Locations (5):
- Y.R.G Ctr, for AIDS Research and Education (11701), Chennai, India
- University of North Carolina Lilongwe CRS (12001), Lilongwe, Malawi
- Wits HIV CRS (11101), Johannesburg, Gauteng, South Africa
- Kilimanjaro Christian Medical CRS, Moshi, Tanzania
- Chiang Mai University ACTG CRS (11501), Chiang Mai, Thailand

REFERENCES:
- [Background] Arribas JR, Pulido F, Delgado R, Lorenzo A, Miralles P, Arranz A, Gonzalez-Garcia JJ, Cepeda C, Hervas R, Pano JR, Gaya F, Carcas A, Montes ML, Costa JR, Pena JM. Lopinavir/ritonavir as single-drug therapy for maintenance of HIV-1 viral suppression: 48-week results of a randomized, controlled, open-label, proof-of-concept pilot clinical trial (OK Study). J Acquir Immune Defic Syndr. 2005 Nov 1;40(3):280-7. doi: 10.1097/01.qai.0000180077.59159.f4. PMID 16249701
- [Background] Campo RE, Lalanne R, Tanner TJ, Jayaweera DT, Rodriguez AE, Fontaine L, Kolber MA. Lopinavir/ritonavir maintenance monotherapy after successful viral suppression with standard highly active antiretroviral therapy in HIV-1-infected patients. AIDS. 2005 Mar 4;19(4):447-9. doi: 10.1097/01.aids.0000161777.38438.ed. No abstract available. PMID 15750401
- [Background] Joly V, Descamps D, Peytavin G, Touati F, Mentre F, Duval X, Delarue S, Yeni P, Brun-Vezinet F. Evolution of human immunodeficiency virus type 1 (HIV-1) resistance mutations in nonnucleoside reverse transcriptase inhibitors (NNRTIs) in HIV-1-infected patients switched to antiretroviral therapy without NNRTIs. Antimicrob Agents Chemother. 2004 Jan;48(1):172-5. doi: 10.1128/AAC.48.1.172-175.2004. PMID 14693536
- [Result] Bartlett JA, Ribaudo HJ, Wallis CL, Aga E, Katzenstein DA, Stevens WS, Norton MR, Klingman KL, Hosseinipour MC, Crump JA, Supparatpinyo K, Badal-Faesen S, Kallungal BA, Kumarasamy N. Lopinavir/ritonavir monotherapy after virologic failure of first-line antiretroviral therapy in resource-limited settings. AIDS. 2012 Jul 17;26(11):1345-54. doi: 10.1097/QAD.0b013e328353b066. PMID 22441252
- [Derived] Kumarasamy N, Aga E, Ribaudo HJ, Wallis CL, Katzenstein DA, Stevens WS, Norton MR, Klingman KL, Hosseinipour MC, Crump JA, Supparatpinyo K, Badal-Faesen S, Bartlett JA. Lopinavir/Ritonavir Monotherapy as Second-line Antiretroviral Treatment in Resource-Limited Settings: Week 104 Analysis of AIDS Clinical Trials Group (ACTG) A5230. Clin Infect Dis. 2015 May 15;60(10):1552-8. doi: 10.1093/cid/civ109. Epub 2015 Feb 18. PMID 25694653

RESULTS

PARTICIPANT FLOW:
Groups:
- LPV/r Monotherapy: Participants will receive lopinavir/ritonavir twice daily for up to 104 weeks. Upon confirmation of virologic failure, emtricitabine (FTC)/tenofovir (TDF) once a day will be added to their regimen.
Period: Screening
Arm/Group | LPV/r Monotherapy
Started | 207 (The number of participants who started this period, is the number of participants who screened.)
Completed | 123 (The number of participants who completed this period, is the number of participants who enrolled.)
Not Completed | 84
Not completed — Did not meet eligibility criteria | 84
Period: Weeks 0 to 24
Arm/Group | LPV/r Monotherapy
Started | 123
Completed | 122 (One subject died prior to week 24.)
Not Completed | 1
Not completed — Death | 1
Period: Weeks 24 to 104
Arm/Group | LPV/r Monotherapy
Started | 122
Completed | 117
Not Completed | 5
Not completed — Death | 3
Not completed — Not able to get to clinic | 2

BASELINE CHARACTERISTICS:
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 123
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 53
Region of Enrollment [Number; unit: participants]
  South Africa | 22
  Thailand | 24
  India | 12
  Malawi | 40
  Tanzania | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Enrolled Participants With Virologic Success at Week 24 on LPV/r Monotherapy
Description: Virologic success at week 24 on LPV/r monotherapy was defined as remaining on LPV/r monotherapy at week 24 without prior virologic failure. Virologic failure was met with either of these two conditions: (i) failure to suppress HIV-1 RNA to < 400 copies/mL by week 24 or (ii) confirmed HIV-1 RNA >= 400 copies/mL after confirmed HIV-1 RNA < 400 copies/mL.
Time Frame: From study entry to week 24
Population: All enrolled individuals.
Measure: Number (90% Confidence Interval); unit: percentage of enrolled subjects
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
percentage of enrolled subjects | 87 [81 to 92]
Statistical Analysis 1: Comparison: LPV/r Monotherapy; The null hypothesis was that LPV/r monotherapy provides at least a 65% short-term virologic response. The target sample size was 120 subjects. Assuming an underlying true 24 week success rate of 76%, this sample size was chosen in order to provide at least 90% power to show that the true 24 week virologic success rate of LPV/r monotherapy in this population is greater than 65%; Test type: Non-Inferiority or Equivalence — Success of the strategy is assessed according to whether the lower bound of the exact 90% confidence interval of this proportion is greater than 65%; confidence interval; Success was determined by whether the lower bound of the 90% exact confidence interval was greater than 65%; proportion = 87, 90% CI 2-sided [81 to 92] — exact confidence interval

2. Primary Outcome: Probability of Grade 3 or 4 Sign or Symptom, or Laboratory Toxicity Over 24 Weeks on Study.
Description: Probability of Grade 3 or 4 sign or symptom, or laboratory toxicity over 24 weeks on study using Kaplan-Meier estimates of the cumulative probability of Grade 3 or 4 sign or symptom, or laboratory toxicity at week 24. Grading of adverse events (signs and symptoms and laboratory toxicities) was according to Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004.
Time Frame: From study entry to week 24
Population: All enrolled individuals.
Measure: Number (95% Confidence Interval); unit: cumulative probability of grade 3 or 4
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
cumulative probability of grade 3 or 4 | 0.23 [0.16 to 0.31]

3. Secondary Outcome: Number of Screened Subjects With at Least One NNRTI, or NRTI-associated Resistance Mutation at A5230 Screening.
Description: Number of screened subjects with at least one NNRTI, or NRTI-associated resistance mutation. Resistance interpretations used the November 30, 2011 Stanford algorithm.
Time Frame: Screening
Population: All screened individuals.
Measure: Number; unit: number of screened subjects
Groups:
- All Screened Subjects With Available Sequences: All screened individuals, for whom a sequence could be obtained, regardless of whether they enrolled or not.
Arm/Group | All Screened Subjects With Available Sequences
Number analyzed (Participants) | 207
number of screened subjects
  At least one NNRTI-associated mutation | 201
  At least one NRTI-associated mutation | 197

4. Secondary Outcome: Time to Treatment Failure, Defined as the First Occurrence of Death, Disease Progression, or Virologic Failure.
Description: 25th percentile in weeks from study entry to treatment failure, defined as the first occurrence of death, disease progression, or virologic failure. Virologic failure was defined as HIV-1 >= 400 copies/mL after week 24 or 2 consecutive HIV-1 RNA >= 400 copies/mL after week 16 following suppression on LPV/r monotherapy.
Time Frame: Study entry to Week 104
Population: All participants enrolled.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
weeks | 48.0 [40.0 to 80.0]

5. Secondary Outcome: Number of Participants With Study-targeted Diagnoses and Clinical Events
Description: Cardiac disorders, Infections and infestations, Metabolism and nutrition disorders, Neoplasms benign, malignant and unspecified (including cysts and polyps), Pregnancy, puerperium and perinatal conditions, Vascular disorders, were specified a priori as study-targeted events by the study chair.
Time Frame: Study entry to week 104
Population: All participants enrolled.
Measure: Number; unit: participants
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
participants | 39

6. Secondary Outcome: Number of Subjects With at Least One New PI-associated Resistance Mutation at Time of Virologic Failure.
Description: Number of subjects with at least one new PI-associated resistance mutation at time of virologic failure. Resistance interpretations used the May 6, 2009 Stanford algorithm.
Time Frame: At time of virologic failure
Population: 16 subjects met the criteria for endpoint failure; 15 subjects were virologic failures and 1 subject intensified prior to virologic failure. Of the 15 subjects with virologic failure, 11 had sequence data, and sequencing failed for 4.
Measure: Number; unit: participants
Groups:
- Virologic Failures by Week 24.: Subjects who met virologic failure criteria by week 24, for whom a sequence could be obtained.
Arm/Group | Virologic Failures by Week 24.
Number analyzed (Participants) | 11
participants | 2

7. Secondary Outcome: Percentage of Subjects Reporting Not Skipping Medications in the Last Month.
Description: The percentage of subjects reporting never missing medications in the last month.
Time Frame: Study entry and weeks 2, 4, 8, 12, 16, 20, and 24
Population: All participants enrolled.
Measure: Number; unit: percentage of subjects with data
Groups:
- LPV/r Monotherapy: Participants will receive lopinavir/ritonavir twice daily for up to 104 weeks. Upon confirmation of virologic failure, emtricitabine (FTC)/tenofovir (TDF) once a day will be added to their regimen. The study is ongoing. Results from entry to week 24 are posted. They will be updated upon completion of study duration of 104 weeks.
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
percentage of subjects with data
  week 2 (N=120) | 90
  week 4 (N=121) | 86.8
  week 8 (N=123) | 87.8
  week 12 (N=123) | 86.2
  week 16 (N=122) | 86.1
  week 20 (N=120) | 90.9
  week 24 (N=122) | 89.4

8. Secondary Outcome: Time to First New Grade 3 or 4 Sign or Symptom or Laboratory Toxicity Following LPV/r Intensification
Description: 25th percentile in weeks from study entry to first new grade 3 or 4 sign or symptom or laboratory toxicity following LPV/r intensification. Grading of adverse events (signs and symptoms and laboratory toxicities) was according to Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004.
Time Frame: From LPV/r intensification to week 104
Population: All participants enrolled.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
weeks | 26.0 [13.1 to 53.3]

9. Secondary Outcome: Level of HIV-1 RNA as Ascertained From Paired DBS and Plasma
Description: Proportion of DBS samples with HIV-1 RNA level <= 400 copies/mL, proportion of plasma samples with HIV-1 RNA level <= 400 copies/mL and proportion of paired DBS and plasma samples that are concordant (both <= 400 copies/mL or both > 400 copies/mL). Results are pooled over 4 different storage temperature conditions (-80C, -20C, 4C and room temperature).
Time Frame: At study entry and weeks 24 and 48
Population: Participants with DBS samples available at study entry, week 24 or 48, with corresponding plasma HIV-1 RNA levels.
Measure: Number; unit: proportion of samples
Units Other Than Participants: paired DBS and plasma samples
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 45
Number analyzed (paired DBS and plasma samples) | 140
proportion of samples
  study entry DBS <= 400 cp/mL | 0.17
  study entry plasma <= 400 cp/mL | 0.00
  study entry DBS & plasma concordance | 0.83
  week 24 DBS <= 400 cp/mL | 0.82
  week 24 plasma <= 400 cp/mL | 0.80
  week 24 DBS & plasma concordance | 0.80
  week 48 DBS <= 400 cp/mL | 0.94
  week 48 plasma <= 400 cp/mL | 0.91
  week 48 DBS & plasma concordance | 0.97

10. Secondary Outcome: HIV-1 Viral Sequence as Ascertained From Paired DBS and Plasma
Description: HIV-1 viral sequencing as ascertained from paired DBS and plasma
Time Frame: At study entry and virologic failure
Population: HIV-1 viral sequence testing in DBS was not performed
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 0

11. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA Levels < 400 Copies/mL From Baseline to Week 104
Time Frame: At Weeks 0, 12, 16, 20, 24, 32, 40, 48, 56, 68, 80, 92, 104
Population: All participants enrolled.
Measure: Number; unit: proportion of participants
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
proportion of participants
  week 0 (N=123) | 0.02
  week 12 (N=122) | 0.75
  week 16 (N=121) | 0.87
  week 20 (N=115) | 0.84
  week 24 (N=122) | 0.84
  week 32 (N=121) | 0.83
  week 40 (N=118) | 0.84
  week 48 (N=118) | 0.87
  week 56 (N=120) | 0.86
  week 68 (N=116) | 0.91
  week 80 (N=117) | 0.85
  week 92 (N=116) | 0.87
  week 104 (N=117) | 0.89

12. Secondary Outcome: Change in CD4+ Cell Counts From Study Entry to Week 104
Time Frame: Study entry and week 104
Population: All participants enrolled.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | LPV/r Monotherapy
Number analyzed (Participants) | 123
cells/mm^3 | 213 [111 to 326]

ADVERSE EVENTS:
Time Frame: From study entry up to 104 weeks.
Description: The protocol required reporting of all signs, symptoms and laboratory abnormalities >= grade 3 and any that led to a study treatment change, regardless of grade. The "DAIDS Table for Grading the Severity of Adult and Pediatric Aes", V1.0, 12/2004 was used.
Groups:
- LPV/r: Participants will receive lopinavir/ritonavir twice daily for up to 104 weeks. Upon confirmation of virologic failure, emtricitabine (FTC)/tenofovir (TDF) once a day will be added to their regimen.
Arm/Group | LPV/r
Serious Adverse Events (participants affected / at risk) | 20/123
Other Adverse Events (participants affected / at risk) | 122/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r (N=123)
Acute myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Gastroenteritis (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 1
Blood cholesterol increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Diabetes mellitus management (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r (N=123)
Abdominal pain (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 12
Chest pain (General disorders) | 13
Pain (General disorders) | 9
Pyrexia (General disorders) | 27
Malaria (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 8
Pneumonia bacterial (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 22
Urinary tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 18
Blood albumin decreased (Investigations) | 22
Blood alkaline phosphatase increased (Investigations) | 10
Blood bicarbonate decreased (Investigations) | 24
Blood bilirubin increased (Investigations) | 7
Blood cholesterol increased (Investigations) | 76
Blood glucose decreased (Investigations) | 9
Blood glucose increased (Investigations) | 31
Blood phosphorus decreased (Investigations) | 39
Blood potassium decreased (Investigations) | 18
Blood sodium decreased (Investigations) | 62
Blood triglycerides increased (Investigations) | 22
Haemoglobin decreased (Investigations) | 15
Low density lipoprotein increased (Investigations) | 54
Neutrophil count decreased (Investigations) | 38
Platelet count decreased (Investigations) | 10
White blood cell count decreased (Investigations) | 19
Headache (Nervous system disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 34
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.